CLINICAL TRIAL: NCT00679939
Title: A 52 Week Randomized, Double-Blind, Multicenter, Mechanistic Study With a 24 Week Open-Label Follow-Up to Evaluate the Effect of AVANDIA TM on Bone in Postmenopausal Women With Type 2 Diabetes Mellitus
Brief Title: Study In Postmenopausal Women With Type 2 Diabetes Looking At Approved Diabetes Drugs And How They Affect Bone Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVD111179
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; bone; x-ray absorptiometry; bone biomarkers; dual-energy; bone mineral density
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Treatment A (Active Comparator): rosiglitazone up to 8mg/day
  Interventions: Drug: Rosiglitazone
- Arm 2 Treatment B (Active Comparator): metformin up to 2000mg/day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Rosiglitazone — up to 8mg/day
  Arms: Arm 1 Treatment A
Drug: Metformin — up to 2000mg/day
  Arms: Arm 2 Treatment B

SUMMARY:
The purpose of this study is to determine the effects of rosiglitazone on the bone in postmenopausal women with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Female, >55 to <80 years
* >5 years menopausal
* Type 2 Diabetes Mellitus (T2DM) diagnosis according to American Diabetes Association (ADA), American Association of Clinical Endocrinologists (AACE), Canadian Diabetes Association (CDA), World Health Organization/International Diabetes Federation (WHO/IDF)
* Drug-naïve (HbA1c < or = 9.0%); OR Prior monotherapy, submaximal doses of metformin (< or = 1000mg Metformin), sulfonylureas (< or = 5mg Glyburide, < or = 10mg Glipizide or < or = 8mg glimepiride) or full dose Januvia (100mg) (HbA1c < or = 8.5%); OR Prior monotherapy, > submaximal doses of metformin (>1000mg) or sulfonylureas (>5mg Glyburide, >10mg Glipizide or >8mg glimepiride) (HbA1c < or = 7.0%)
* Weighs <300 lbs (136.4 kg)
* Two or more vertebra (L1-L4) suitable for BMD measurement by dual x-ray absorptiometry (DXA)
* Absolute BMD value consistent with T-score >-2.5 at femoral neck, lumbar spine and total hip

Exclusion Criteria:

* Type 1 Diabetes Mellitus (T1DM) or history of diabetic ketoacidosis (DKA)
* Renal or hepatic disease (clinically significant)
* Hepatocellular reaction, severe edema, or medically serious fluid event associated with thiazolidinedione (TZD)
* Recent (<6mos) history or clinical intervention for angina or myocardial infarction or is taking nitrates
* Any stage of heart failure, i.e. New York Heart Association (NYHA) class I-IV
* Systolic BP >160mmHg or diastolic BP >90mmHg while on antihypertensive
* Hypersensitivity to TZDs, biguanides
* Prior treatment with two or more oral anti-diabetic (OAD) agents
* Bilateral hip replacements
* Concurrent diseases affecting bone metabolism
* Active malabsorption syndrome
* Serum calcium outside the central lab reference range
* Thyroid replacement therapy, serum thyroid stimulating hormone (TSH) must be within range
* Vitamin D deficiency
* Previous treatment with: strontium, intravenous (IV) bisphosphonate, fluoride, hormones, calcineurin inhibitors or methotrexate
* Chronic systemic corticosteroid [e.g. glucocorticoid, mineralocorticoid] treatment of no more than two intra-articular injections within the past year or use of oral parenteral, or long-term, high-dose inhaled corticosteroids

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2008-04-21; Primary Completion 2010-09-16 (Actual); Study Completion 2010-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (18):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Wenatchee, Washington
- Argentina (2):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Granby, Quebec
- GSK Investigational Site, Tallinn, Estonia
- Mexico (4):
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Durango
- GSK Investigational Site, Lahore, Pakistan
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marikina City
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Benidorm/Alicante
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Petrel

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Fitzpatrick LA, Bilezikian JP, Wooddell M, Paul G, Kolatkar NS, Nino AJ, Miller CG, Bogado CE, Arnaud CD, Cobitz AR. Mechanism of action study to evaluate the effect of rosiglitazone on bone in postmenopausal women with type 2 diabetes mellitus: rationale, study design and baseline characteristics. J Drug Assess. 2011 Dec 16;1(1):11-9. doi: 10.3109/21556660.2011.641703. eCollection 2012. PMID 27536422
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Miller CG, Bogado CC, Nino AJ, Northcutt AR, Yu HJ, Lewiecki EM, Paul G, Cobitz AR, Wooddell MJ, Bilezikian JP, Fitzpatrick LA. Evaluation of Quantitative Computed Tomography Cortical Hip Quadrant in a Clinical Trial With Rosiglitazone: A Potential New Study Endpoint. J Clin Densitom. 2016 Oct;19(4):485-491. doi: 10.1016/j.jocd.2016.02.003. Epub 2016 Mar 24. PMID 27052635
- [Derived] Bilezikian JP, Josse RG, Eastell R, Lewiecki EM, Miller CG, Wooddell M, Northcutt AR, Kravitz BG, Paul G, Cobitz AR, Nino AJ, Fitzpatrick LA. Rosiglitazone decreases bone mineral density and increases bone turnover in postmenopausal women with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2013 Apr;98(4):1519-28. doi: 10.1210/jc.2012-4018. Epub 2013 Feb 28. PMID 23450056
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVD111179 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosiglitazone in DB Period; Metformin in OL Period: Rosiglitazone (RSG) initiated at a total daily dose of 4 milligrams (mg) in the 52-week DB Period. RSG could be uptitrated to a total daily dose of 8 mg at Week 4. At Week 52, all participants were switched to open-label (OL) Metformin (MET) therapy for 24 weeks during the follow-up phase; all participants were force-titrated from 1000 mg/day to 2000 mg/day over a 4-week period. However, participants could be down-titrated to alleviate any MET-related tolerability issues.
- Metformin in DB Period; Metformin in OL Period: Metformin (MET) initiated at a total daily dose of 1000 mg in the 52-week DB Period. MET could be uptitrated to 1500 mg/day at Week 2 and to 2000 mg/day at Week 4. At Week 52, all participants were switched to open-label MET therapy for 24 weeks during the follow-up phase; all participants were force-titrated from 1000 mg/day to 2000 mg/day over a 4-week period. However, participants could be down-titrated to alleviate any MET-related tolerability issues.
Period: 52-Week Double-Blind (DB) Period
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Started | 114 | 112
Completed | 77 | 85
Not Completed | 37 | 27
Not completed — Withdrew Consent | 17 | 13
Not completed — Adverse Event | 14 | 12
Not completed — Investigator Discretion | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Period: 24-Week Open-Label (OL) Period
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Started | 76 (One participant who completed the DB Period did not receive the OL dose of MET.) | 84 (One participant who completed the DB Period did not receive the OL dose of MET.)
Completed | 69 | 80
Not Completed | 7 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Met Stopping Criteria | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period | Total
Number analyzed (Participants) | 114 | 111 | 225
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristics were summarized for all participants in the Safety Population, comprised of all randomized participants who received at least one dose of study medication. One participant in the Metformin arm did not receive study medication and was not included in the Safety Population.
  Years | 63.6 (6.61) | 64.0 (6.46) | 63.8 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristics were summarized for all participants in the Safety Population, comprised of all randomized participants who received at least one dose of study medication. One participant in the Metformin arm did not receive study medication and was not included in the Safety Population.
  Participants
    Female | 114 | 111 | 225
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Baseline Characteristics were summarized for all participants in the Safety Population, comprised of all randomized participants who received at least one dose of study medication. One participant in the Metformin arm did not receive study medication and was not included in the Safety Population.
  participants
    White - White/Caucasian/European | 82 | 78 | 160
    African American/African | 2 | 8 | 10
    American Indian or Alaskan Native | 6 | 5 | 11
    Asian - Central/South Asian | 13 | 10 | 23
    South East Asian | 4 | 6 | 10
    Mixed Race | 3 | 2 | 5
    East Asia | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Bone Mineral Density (BMD) Via Dual-energy X-ray Absorptiometry (DXA) at Week 52
Description: FN BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Bone mineral density is calculated as the mineral content of a bone divided by the area of the bone. DXA is the principal technique used for measuring BMD. Percent change from Baseline at Week 52 was calculated as (BMD at Week 52 minus BMD at Baseline)/BMD at Baseline x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Change in FN BMD at Week 52 was only analyzed within the Rosiglitazone arm.
Time Frame: Baseline and Week 52
Population: Safety Population. Only evaluable participants with a value at baseline and at Week 52 for the parameter of interest were analyzed. Only participants with Baseline DXA and Week 52 DXA measurements performed on or prior to initiating open-label MET are included in this primary analysis.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period
Number analyzed (Participants) | 52
percent change | -1.24 (0.619)

2. Primary Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Bone Mineral Density (BMD) Via Dual-energy X-ray Absorptiometry (DXA) at Week 76+10 Days
Description: FN BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Bone mineral density is calculated as the mineral content of a bone divided by the area of the bone. DXA is the principal technique used for measuring BMD. Percent change from Baseline at Week 76+10 days was calculated as (BMD at Week 76+10 days minus BMD at Baseline)/BMD at Baseline x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline and Week 76+10 days
Population: Safety Population. Only evaluable participants with a value at baseline and at Week 76 performed up to 10 days after stopping OL MET for the parameter of interest were analyzed.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 65 | 70
percent change | -1.91 (0.624) | 0.31 (0.636)

3. Primary Outcome: Adjusted Percent Change in Femoral Neck (FN) Bone Mineral Density (BMD) Via Dual-energy X-ray Absorptiometry (DXA) From Week 52 +10 Days to Week 76+10 Days
Description: FN BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Bone mineral density is calculated as the mineral content of a bone divided by the area of the bone. DXA is the principal technique used for measuring BMD. Percent change from Week 52+10 days to Week 76+10 days was calculated as (BMD at Week 76+10 days minus BMD at Week 52+10 days)/BMD at Week 52+10 days x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52+10 days and Week 76+10 days
Population: Safety Population. Only evaluable participants with a value at Week 52 performed up to 10 days after initiating OL MET and at Week 76 performed up to 10 days after stopping OL MET for the parameter of interest were analyzed.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 56 | 62
percent change | -0.07 (0.589) | -0.02 (0.585)

4. Secondary Outcome: Adjusted Percent Change From Baseline in Femoral Neck, Total Hip, Trochanter, and Lumbar Spine BMD Via DXA at Week 52
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Percent change from Baseline at Week 52 was calculated as (BMD at Week 52 minus BMD at Baseline)/BMD at Baseline x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline and Week 52
Population: Safety Population. Only evaluable participants with a value at baseline and at Week 52 for the parameter of interest were analyzed. Only participants with Baseline DXA and Week 52 DXA measurements performed on or prior to initiating open-label MET were analyzed. Not all participants had correct positioning for the DXA lumbar spine measurement.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 52 | 54
percent change
  Femoral neck, n=52, 54 | -1.24 (0.619) | 0.72 (0.659)
  Total hip, n=52, 54 | -0.77 (0.417) | -0.38 (0.440)
  Trochanter, n=52, 54 | -0.21 (0.725) | -0.78 (0.768)
  Lumbar spine, n=51, 53 | -1.21 (0.473) | 0.12 (0.505)

5. Secondary Outcome: Adjusted Percent Change in Femoral Neck, Total Hip, Trochanter, and Lumbar Spine BMD Via DXA From Week 52+10 Days to Week 76 + 10 Days
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Percent change from Week 52 + 10 days toat Week 76 + 10 days was calculated as (BMD at Week 76 + 10 days minus BMD at Week 52 + 10 days)/BMD at Week 52 + 10 days x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 + 10 days and Week 76 + 10 days
Population: Safety Population. Only evaluable participants with a value at Week 52 performed up to 10 days after initiating OL MET and at Week 76 performed up to 10 days after stopping OL MET for the parameter of interest were analyzed. Not all participants had correct positioning for the DXA lumbar spine measurement.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 56 | 62
percent change
  Femoral neck, n=56, 62 | -0.07 (0.589) | -0.02 (0.585)
  Total hip, n=56, 62 | 0.40 (0.304) | -0.13 (0.301)
  Trochanter, n=56, 62 | -0.02 (0.475) | -0.68 (0.469)
  Lumbar spine, n=55, 62 | 0.26 (0.440) | 1.03 (0.442)

6. Secondary Outcome: Adjusted Percent Change in Femoral Neck, Total Hip, Trochanter, and Lumbar Spine BMD Via DXA From Week 52+30 Days to Week 76 + 30 Days
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (BMD at Week 76 + 30 days minus BMD at Week 52 + 30 days)/BMD at Week 52 + 30 days x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: Safety Population. Only evaluable participants with a value at Week 52 performed up to 30 days after initiating OL MET and Week 76 performed up to 30 days after stopping OL MET for the parameter of interest were analyzed. Not all participants had correct positioning for all of the DXA measurements.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 65 | 73
percent change
  Femoral neck, n=64, 73 | -0.27 (0.559) | -0.25 (0.535)
  Total hip, n=64, 73 | 0.00 (0.298) | -0.27 (0.283)
  Trochanter, n=64, 73 | -0.17 (0.495) | -0.47 (0.470)
  Lumbar spine, n=65, 70 | 0.54 (0.445) | 0.90 (0.442)

7. Secondary Outcome: Adjusted Percent Change From Baseline in Bone Specific Alkaline Phosphatase (BSAP) and Procollagen Type 1 N-propeptide (P1NP) at Week 52 and Week 76
Description: BSAP and P1NP levels were measured in micrograms per liter (mcg/L) from blood samples. BSAP and P1NP are indicators of bone buildup or formation. GM, geometric mean; SE, standard error. Percent change was based on log-transformed data and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52, and Week 76
Population: Safety Population. Only evaluable participants with a value at Baseline and at Week 52 or Week 76 for the parameter of interest were analyzed.
Measure: Number; unit: percent change
Groups:
- Rosiglitazone: Rosiglitazone (RSG) initiated at a total daily dose of 4 milligrams (mg). RSG could be uptitrated to a total daily dose of 8 mg at Week 4. At Week 52, all participants were switched to open-label Metformin (MET) therapy for 24 weeks during the follow-up phase; all participants were force-titrated from 1000 mg/day to 2000 mg/day over a 4-week period. However, participants could be down-titrated to alleviate any MET-related tolerability issues.
- Metformin: Metformin (MET) initiated at a total daily dose of 1000 mg. MET could be uptitrated to 1500 mg/day at Week 2 and to 2000 mg/day at Week 4. At Week 52, all participants were switched to open-label MET therapy for 24 weeks during the follow-up phase; all participants were force-titrated from 1000 mg/day to 2000 mg/day over a 4-week period. However, participants could be down-titrated to alleviate any MET-related tolerability issues.
Arm/Group | Rosiglitazone | Metformin
Number analyzed (Participants) | 78 | 84
percent change
  Week 52, GM - SE, BSAP, n=78, 84 | -15.2 | -29.7
  Week 52, GM, BSAP, n=78, 84 | -12.3 | -27.3
  Week 52, GM + SE, BSAP, n=78, 84 | -9.3 | -24.8
  Week 76, GM - SE, BSAP, n=64, 77 | -18.7 | -26.7
  Week 76, GM, BSAP, n=64, 77 | -15.9 | -24.3
  Week 76, GM + SE, BSAP, n=64, 77 | -12.9 | -21.8
  Week 52, GM - SE, P1NP, n=76, 83 | 5.0 | -16.5
  Week 52, GM, P1NP, n=76, 83 | 9.0 | -13.3
  Week 52, GM + SE, P1NP, n=76, 83 | 13.3 | -9.9
  Week 76 GM - SE, P1NP, n=63, 75 | -11.2 | -14.5
  Week 76, GM, P1NP, n=63, 75 | -6.9 | -10.5
  Week 76, GM + SE, P1NP, n=63, 75 | -2.4 | -6.4

8. Secondary Outcome: Adjusted Percent Change in Bone Specific Alkaline Phosphatase (BSAP) and Procollagen Type 1 N-propeptide (P1NP) From Week 52 to Week 76
Description: as for outcome 7
Time Frame: Week 52 and Week 76
Population: Safety Population. Only evaluable participants with a value at Week 52 and at Week 76 for the parameter of interest were analyzed. One participant did not have P1NP measured.
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 76
percent change
  GM - SE, BSAP, n=64, 76 | -5.6 | 4.3
  GM, BSAP, n=64, 76 | -2.0 | 8.0
  GM + SE, BSAP, n=64, 76 | 1.8 | 11.8
  GM - SE, P1NP, n=63, 76 | -15.8 | 3.2
  GM, P1NP, n=63, 76 | -12.4 | 7.0
  GM + SE, P1NP, n=63, 76 | -9.0 | 11.0

9. Secondary Outcome: Adjusted Percent Change From Baseline in Carboxyterminal Cross-linked Telopeptide of Type 1 Collagen (CTX) at Week 52 and Week 76
Description: CTX levels were measured in picograms per milliliter (pg/ml) from blood samples. CTX is an indicator of bone break down or resorption. Percent change was based on log-transformed data and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 77 | 84
percent change
  Week 52, GM - SE, n=77, 84 | 11.3 | -7.8
  Week 52, GM, n=77, 84 | 18.1 | -2.3
  Week 52, GM + SE, n=77, 84 | 25.4 | 3.7
  Week 76, GM - SE, n=63, 77 | -19.5 | -4.5
  Week 76, GM, n=63, 77 | -13.1 | 2.6
  Week 76, GM + SE, n=63, 77 | -6.1 | 10.3

10. Secondary Outcome: Adjusted Percent Change in Carboxyterminal Cross-linked Telopeptide of Type 1 Collagen (CTX) From Week 52 to Week 76
Description: as for outcome 9
Time Frame: Week 52 and Week 76
Population: Safety Population. Only evaluable participants with a value at Week 52 and at Week 76 for the parameter of interest were analyzed.
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 76
percent change
  GM - SE | -31.2 | 2.2
  GM | -26.7 | 8.4
  GM + SE | -21.9 | 14.9

11. Secondary Outcome: Adjusted Percent Change From Baseline in 25-Hydroxyvitamin D (Vitamin D) at Week 52 and Week 76
Description: Vitamin D levels were measured in nanomoles per Liter (nmol/L) from blood samples. Vitamin D is required for good bone health. Percent change was based on log-transformed data and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 61 | 65
percent change
  Week 52, GM - SE, n=61, 65 | -27.9 | -15.9
  Week 52, GM, n=61, 65 | -24.7 | -12.2
  Week 52, GM + SE, n=61, 65 | -21.4 | -8.4
  Week 76, GM - SE, n=55, 58 | -21.3 | -12.5
  Week 76, GM, n=55, 58 | -18.1 | -8.9
  Week 76, GM + SE, n=55, 58 | -14.6 | -5.2

12. Secondary Outcome: Adjusted Percent Change in 25-Hydroxyvitamin D (Vitamin D) From Week 52 to Week 76
Description: as for outcome 11
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 63 | 76
percent change
  GM - SE | -4.7 | -7.7
  GM | 0.1 | -3.2
  GM + SE | 5.1 | 1.5

13. Secondary Outcome: Adjusted Percent Change From Baseline in Intact Parathyroid Hormone (PTH) at Week 52 and Week 76
Description: Intact PTH levels were measured in nanograms per Liter (ng/L) from blood samples. Intact PTH is the amount of PTH circulating in the blood and influences bone health. Percent change was based on log-transformed data and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 71
percent change
  Week 52, GM - SE, n=64, 71 | -16.5 | -25.9
  Week 52, GM, n=64, 71 | -12.0 | -22.0
  Week 52, GM + SE, n=64, 71 | -7.2 | -17.8
  Week 76, GM - SE, n=56, 64 | -28.8 | -26.2
  Week 76, GM, n=56, 64 | -23.1 | -20.8
  Week 76, GM + SE, n=56, 64 | -17.0 | -15.0

14. Secondary Outcome: Adjusted Percent Change in Intact Parathyroid Hormone (PTH) From Week 52 to Week 76
Description: as for outcome 13
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 75
percent change
  GM - SE | -13.2 | -1.7
  GM | -7.4 | 4.3
  GM + SE | -1.3 | 10.7

15. Secondary Outcome: Percent Change From Baseline in Serum Estradiol at Week 52 and Week 76
Description: Serum estradiol levels were measured in picomoles per Liter (pmol/L) from blood samples. Estradiol is one form of the female sex hormone estrogen and influences bone health. Percent change from baseline was based on log-transformed data.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 74 | 82
percent change
  Week 52, GM - SE, n=74, 82 | -17.0838 | -31.4166
  Week 52, GM, n=74, 82 | -3.453 | -17.280
  Weel 52, GM + SE, n=74, 82 | 12.4189 | -0.2292
  Week 76, GM - SE, n=64, 76 | -16.0971 | 0.4372
  Week 76, GM, n=64, 76 | 0.215 | 21.389
  Week 76, GM + SE, n=64, 76 | 19.6987 | 46.7122

16. Secondary Outcome: Percent Change in Serum Estradiol From Week 52 to Week 76
Description: as for outcome 15
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 77
percent change
  GM - SE | -15.2056 | 29.3058
  GM | 0.513 | 50.823
  GM + SE | 19.1447 | 75.9217

17. Secondary Outcome: Percent Change From Baseline in Total Testosterone at Week 52 and Week 76
Description: Total testosterone levels were measured in nanomoles per Liter (nmol/L) from blood samples. Testosterone is a male sex hormone and influences bone health; total testosterone is the entire amount circulating in blood. Percent change from baseline was based on log-transformed data.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 74 | 82
percent change
  Week 52, GM - SE, n=74, 82 | 14.1569 | -5.8206
  Week 52, GM, n=74, 82 | 19.689 | 1.044
  Week 52, GM + SE, n=74, 82 | 25.4897 | 8.4082
  Week 76, GM - SE, n=64, 75 | -12.5441 | -8.2870
  Week 76, GM, n=64, 75 | -8.156 | -2.932
  Week 76, GM + SE, n=64, 75 | -3.5470 | 2.7363

18. Secondary Outcome: Percent Change in Total Testosterone From Week 52 to Week 76
Description: as for outcome 17
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 76
percent change
  GM - SE | -29.0307 | -13.9923
  GM | -24.373 | -7.102
  GM + SE | -19.4104 | 0.3411

19. Secondary Outcome: Percent Change From Baseline in Free Testosterone at Week 52 and Week 76
Description: Free testosterone levels were measured as a percentage of total testosterone from blood samples. Free testosterone is the amount of testosterone available to the body for use. Percent change from baseline was based on log-transformed data.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 74 | 82
percent change
  Week 52, GM - SE, n=74, 82 | -9.9964 | 2.5725
  Week 52, GM, n=74, 82 | -5.940 | 6.266
  Week 52, GM + SE, n=74, 82 | 1.7006 | 10.0934
  Week 76, GM - SE, n=64, 75 | -0.3232 | -1.9532
  Week 76, GM, n=64, 75 | 3.687 | 2.478
  Week 76, GM + SE, n=64, 75 | 7.8593 | 7.1093

20. Secondary Outcome: Percent Change in Free Testosterone From Week 52 to Week 76
Description: as for outcome 19
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 76
percent change
  GM - SE | 3.1109 | -6.9549
  GM | 8.993 | -3.537
  GM + SE | 15.2100 | 0.0073

21. Secondary Outcome: Percent Change From Baseline in Sex Hormone Binding Globulin (SHBG) at Week 52 and Week 76
Description: SHBG levels were measured in nanomoles per liter (nmol/L) from blood samples. SHBG binds to estradiol and testosterone and influences the amount of estradiol or testosterone available to the body for use. Percent change from baseline was based on log-transformed data.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 74 | 83
percent change
  Week 52, GM - SE, n=74, 83 | 33.2608 | 4.3929
  Week 52, GM, n=74, 83 | 37.563 | 8.146
  Week 52, GM + SE, n=74, 83 | 42.0049 | 12.0349
  Week 76, GM - SE, n=61, 67 | -0.2973 | 4.0983
  Week 76, GM, n=61, 67 | 3.137 | 9.846
  Week 76, GM + SE, n=61, 67 | 6.6896 | 15.9116

22. Secondary Outcome: Percent Change in Sex Hormone Binding Globulin (SHBG) From Week 52 to Week 76
Description: as for outcome 21
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 62 | 66
percent change
  GM - SE | -27.0129 | -3.9036
  GM | -24.624 | -0.825
  GM + SE | -22.1566 | 2.3517

23. Other Pre Specified Outcome: Percent Change in Percentage of Free Estradiol From Week 52 to Week 76
Description: Free estradiol levels were measured as a percentage of serum estrogen from blood samples. Free estradiol is the amount of estrogen available to the body for use. Percent change was based on log-transformed data.
Time Frame: Week 52 and Week 76
Population: Safety Population. Only evaluable participants with a value at Week 52 and Week 76 for the parameter of interest were analyzed.
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 33 | 38
percent change
  GM - SE | -7.6337 | -5.4666
  GM | -2.683 | -0.975
  GM + SE | 2.5337 | 3.7301

24. Other Pre Specified Outcome: Percent Change in Free Estradiol From Week 52 to Week 76
Description: Free estradiol levels were measured in picomoles per Liter (pmol/L) from blood samples. Free estrodial is the amount of estrogen available to the body for use. Change was based on log-transformed data.
Time Frame: Week 52 and Week 76
Population: as for outcome 23
Measure: Number; unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 27 | 33
percent change
  GM - SE | -29.5250 | 96.1843
  GM | -3.239 | 173.932
  GM + SE | 32.8525 | 282.4903

25. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck, Total Hip, Trochanter, and Lumbar Spine BMD Via DXA at Week 52 + 10 Days and Week 76 + 10 Days
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Percent change from Baseline at Week 52 + 10 days or Week 76 + 10 days was calculated as (BMD at Week 52 + 10 days (or Week 76 + 10 days ) minus BMD at Baseline)/BMD at Baseline x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 10 days, and Week 76 + 10 days
Population: Safety Population. Only evaluable participants with a value at Baseline and at Week 52 performed up to 10 days after initiating OL MET or at Week 76 performed up to 10 days after stopping OL MET for the parameter of interest were analyzed. Not all participants had the correct positioning for the DXA lumbar spine measurement.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 70 | 78
percent change
  Week 52 + 10 days; Femoral neck (FN), n=70, 78 | -1.47 (0.521) | 0.22 (0.512)
  Week 52 + 10 days; Total hip (TH), n=70, 78 | -1.62 (0.386) | -0.72 (0.379)
  Week 52 + 10 days; Trochanter (Tro.), n=70, 78 | -1.45 (0.602) | -1.04 (0.589)
  Week 52 + 10 days; Lumbar spine (LS), n=70, 76 | -1.41 (0.416) | 0.04 (0.419)
  Week 76 + 10 days; FN, n=65, 70 | -1.91 (0.624) | 0.31 (0.636)
  Week 76 + 10 days; TH, n=65, 70 | -1.70 (0.415) | -0.83 (0.420)
  Week 76 + 10 days; Tro., n=65, 70 | -2.14 (0.644) | -1.35 (0.650)
  Week 76 + 10 days; LS, n=65, 71 | -1.24 (0.452) | 0.85 (0.457)

26. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck, Total Hip, Trochanter, and Lumbar Spine BMD Via DXA at Week 52 + 30 Days and Week 76 + 30 Days
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by DXA. Percent change from Baseline at Week 52 + 30 days or Week 76 + 30 days was calculated as (BMD at Week 52 + 30 days (or Week 76 + 30 days) minus BMD at Baseline)/BMD at Baseline x 100% and was assessed by analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: Safety Population. Only evaluable participants with a value at Baseline and at Week 52 performed up to 30 days after initiating OL MET or at Week 76 performed up to 30 days after stopping OL MET for the parameter of interest were analyzed. Not all participants had the correct positioning for all of the DXA measurements.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 79 | 83
percent change
  Week 52 + 30 days; Femoral neck (FN), n=77, 83 | -1.59 (0.503) | 0.24 (0.498)
  Week 52 + 30 days; Total hip (TH), n=77, 83 | -1.79 (0.370) | -0.72 (0.364)
  Week 52 + 30 days; Trochanter (Tro.), n=77, 83 | -1.83 (0.583) | -1.01 (0.574)
  Week 52 + 30 days; Lumbar spine (LS), n=79, 81 | -1.60 (0.417) | 0.11 (0.421)
  Week 76 + 30 days; FN, n=66, 74 | -2.05 (0.620) | 0.29 (0.619)
  Week 76 + 30 days; TH, n=66, 74 | -1.79 (0.408) | -0.68 (0.404)
  Week 76 + 30 days; Tro., n=66, 74 | -2.53 (0.508) | -0.96 (0.575)
  Week 76 + 30 days; LS, n=66, 72 | -1.15 (0.464) | 1.13 (0.467)

27. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck, Total Hip, Trochanter, and Intertrochanter Areal BMD Via Quantitative Computed Tomography (QCT) at Week 52 + 30 Days and Week 76 + 30 Days
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by QCT. BMD by QCT is the 2-dimensional volume that mimics the DXA measurement for the same region. Percent change from Baseline at Week 52 + 30 days orWeek 76 + 30 days was calculated as (BMD at Week 52 + 30 days (orWeek 76 + 30 days) minus BMD at baseline)/BMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: Safety Population, QCT subset. Only evaluable participants with a value at Baseline and at Week 52 performed up to 30 days after initiating OL MET or at Week 76 performed up to 30 days after stopping OL MET for the parameter of interest were analyzed.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days; Femoral neck (FN), n=32, 35 | -2.39 (0.895) | 0.09 (0.986)
  Week 52 + 30 days; Total hip (TH), n=32, 35 | -3.39 (0.475) | 0.09 (0.521)
  Week 52 + 30 days; Trochanter (Tro.), n=32, 35 | -4.53 (0.612) | -0.23 (0.669)
  Week 52+30 days; Intertrochanter (Inter.),n=32, 35 | -3.36 (0.515) | 0.77 (0.565)
  Week 76+30 days; Femoral neck (FN), n=31, 30 | -1.98 (0.587) | -1.52 (0.705)
  Week 76 + 30 days; TH, n=31, 30 | -2.11 (0.495) | -0.32 (0.591)
  Week 76 + 30 days; Tro., n=31, 30 | -2.86 (0.752) | -1.28 (0.892)
  Week 76 + 30 days; Inter., n=31, 30 | -1.66 (0.525) | 0.30 (0.627)

28. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck, Total Hip, Trochanter, and Intertrochanter Areal BMD Via Quantitative Computed Tomography (QCT) From Week 52+30 Days to Week 76 + 30 Days
Description: BMD (measured in grams per centimeters squared [g/cm^2]) was measured by QCT. BMD by QCT is the 2-dimensional volume that mimics the DXA measurement for the same region. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (BMD at Week 76 + 30 days minus BMD at Week 52 + 30 days)/BMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: Safety Population, QCT subset. Only evaluable participants with a value at Week 52 performed up to 30 days after initiating OL MET or at Week 76 performed up to 30 days after stopping OL MET for the parameter of interest were analyzed.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  percent change | 0.95 (0.728) | -1.39 (0.866)
  Total hip | 1.61 (0.346) | -0.18 (0.411)
  Trochanter | 1.81 (0.534) | -0.91 (0.632)
  Intertrochanter | 2.05 (0.428) | -0.25 (0.507)

29. Post Hoc Outcome: Adjusted Percent Change From Baseline in Total Hip (TH) Integral, TH Trabecular, and TH Cortical vBMD Via QCT at Week 52 + 30 Days and at Week 76 + 30 Days
Description: Volumetric (v)BMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. vBMD is the 3-dimensional density of a region of bone. Cortical bone is dense bone. Trabecular bone is spongy bone. Integral bone is the sum of cortical and trabecular bone measurements. Cortical thickness is the width of the cortical shell. Percent change from Baseline was calculated as (vBMD at Week 52+30 days (or Week 76+30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days; Integral, n=32, 35 | -3.60 (0.587) | 0.99 (0.645)
  Week 52 + 30 days; Trabecular, n=32, 35 | -3.63 (1.243) | 0.21 (1.376)
  Week 52 + 30 days; Cortical, n=32, 35 | -0.54 (0.537) | 0.52 (0.603)
  Week 76 + 30 days; Integral, n=31, 30 | -1.70 (0.657) | 0.85 (0.786)
  Week 76 + 30 days; Trabecular, n=31, 30 | -2.66 (1.211) | 0.70 (1.445)
  Week 76 + 30 days; Cortical, n=31, 30 | 0.23 (0.421) | 0.50 (0.518)

30. Post Hoc Outcome: Adjusted Percent Change in Total Hip (TH) Integral, TH Trabecular, and TH Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: Volumetric (v)BMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. vBMD is the 3-dimensional density of a region of bone. Cortical bone is dense bone. Trabecular bone is spongy bone. Integral bone is the sum of cortical and trabecular bone measurements. Cortical thickness is the width of the cortical shell. Percent change from Week 52 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/ vBMD at Week 52 + 30 days x 100% and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  Integral | 2.24 (0.483) | -0.20 (0.5746)
  Trabecular | 0.90 (1.252) | 1.15 (1.491)
  Cortical | 0.94 (0.449) | -0.06 (0.548)

31. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Integral, FN Trabecular, and FN Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 days or Week 76 + 30 days was calculated as (vBMD at Week 52 + 30 days (orWeek 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -3.72 (1.097) | 0.58 (1.208)
  Week 52 + 30 days, Trabecular, n=32, 35 | -1.83 (1.695) | 0.91 (1.867)
  Week 52 + 30 days, Cortical, n=32, 35 | -1.00 (0.735) | -0.20 (0.819)
  Week 76 + 30 days, Integral, n=31, 30 | -2.13 (0.946) | -0.61 (1.141)
  Week 76 + 30 days, Trabecular, n=31, 30 | -1.05 (1.798) | 2.27 (2.141)
  Week 76 + 30 days, Cortical, n=31, 30 | -0.46 (0.599) | -1.60 (0.723)

32. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Integral, FN Trabecular, and FN Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/vBMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  Integral | 2.21 (0.871) | -1.37 (1.040)
  Trabecular | 0.27 (1.721) | 2.21 (2.044)
  Cortical | 1.03 (0.774) | -1.30 (0.929)

33. Post Hoc Outcome: Adjusted Percent Change From Baseline in Trochanter Integral, Trochanter Trabecular, and Trochanter Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 days or Week 76 + 30 days was calculated as (vBMD at Week 52 + 30 days (or Week 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -4.80 (0.666) | 0.01 (0.730)
  Week 52 + 30 days, Trabecular, n=32, 35 | -3.43 (1.157) | 0.67 (1.275)
  Week 52 + 30 days, Cortical, n=32, 35 | -1.26 (0.490) | -0.18 (0.540)
  Week 76 + 30 days, Integral, n=31, 30 | -2.88 (0.748) | -0.93 (0.889)
  Week 76 + 30 days, Trabecular, n=31, 30 | -2.42 (1.085) | 0.92 (1.293)
  Week 76 + 30 days, Cortical, n=31, 30 | -0.49 (0.384) | -0.64 (0.462)

34. Post Hoc Outcome: Adjusted Percent Change in Trochanter Integral, Trochanter Trabecular, and Trochanter Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: as for outcome 32
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  percent change | 2.22 (0.506) | -0.90 (0.600)
  Trabecular | 1.07 (1.138) | 0.95 (1.353)
  Cortical | 0.78 (0.396) | -0.65 (0.474)

35. Post Hoc Outcome: Adjusted Percent Change From Baseline in Intertrochanter Integral, Intertrochanter Trabecular, and Intertrochanter Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: as for outcome 33
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -3.47 (0.621) | 2.18 (0.683)
  Week 52 + 30 days, Trabecular, n=32, 35 | -4.26 (1.341) | -0.22 (1.485)
  Week 52 + 30 days, Cortical, n=32, 35 | -0.76 (0.568) | 0.99 (0.631)
  Week 76 + 30 days, Integral, n=31, 30 | -0.92 (0.746) | 1.88 (0.895)
  Week 76 + 30 days, Trabecular, n=31, 30 | -3.09 (1.278) | 0.27 (1.525)
  Week 76 + 30 days, Cortical, n=31, 30 | 0.41 (0.472) | 0.79 (0.573)

36. Post Hoc Outcome: Adjusted Percent Change in Intertrochanter Integral, Intertrochanter Trabecular, and Intertrochanter Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: as for outcome 32
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  percent change | 2.83 (0.563) | -0.46 (0.671)
  Trabecular | 1.16 (1.298) | 1.21 (1.545)
  Cortical | 1.29 (0.479) | -0.27 (0.577)

37. Post Hoc Outcome: Adjusted Percent Change From Baseline in Vertebral Trabecular vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: BMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 days or Week 76 + 30 days was calculated as (vBMD at Week 52 + 30 days (orWeek 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, n=32, 35 | -6.71 (1.454) | -1.72 (1.601)
  Week 76 + 30 days, n=31, 30 | -5.15 (1.121) | -3.91 (1.337)

38. Post Hoc Outcome: Adjusted Percent Change in Vertebral Trabecular vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: BMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/vBMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change | 3.53 (1.454) | -2.11 (1.727)

39. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Supero-posterior Integral, Trabecular, and Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 days orWeek 76 + 30 days was calculated as (vBMD at Week 52 + 30 days (or Week 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therpay, and region. Supero-posterior is the upper and back section of the FN.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: Safety Population, QCT subset. Only evaluable participants with a value at Baseline and at Week 52 performed up to 30 days after initiating OL MET or Week 76 performed up to 30 days after stopping OL MET for the parameter of interest were analyzed.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -10.26 (2.194) | -0.03 (2.417)
  Week 52 + 30 days, Trabecular, n=32, 35 | 2.77 (5.848) | 5.57 (6.420)
  Week 52 + 30 days, Cortical, n=32, 35 | -3.76 (0.836) | -0.66 (0.922)
  Week 76 + 30 days, Integral, n=31, 30 | -4.21 (2.094) | 1.07 (2.508)
  Week 76 + 30 days, Trabecular, n=31, 30 | 2.37 (7.040) | 10.24 (8.362)
  Week 76 + 30 days, Cortical, n=31, 30 | -1.65 (0.730) | -1.30 (0.877)

40. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Supero-posterior and Cortical vBMD Via QCT at Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Baseline at Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at baseline and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Supero-posterior is the upper and back section of the FN.
Time Frame: Baseline and Week 76 + 30 days
Population: Safety Population, QCT subset. Only evaluable participants with a value at Baseline and at Week 76 performed up to 30 days after stopping OL MET for the parameter of interest were analyzed.
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
mg/cm^3 | -8.007 (3.4199) | -7.006 (4.1114)

41. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Supero-posterior Integral, Trabecular, and Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/vBMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therpay, and region. Supero-posterior is the upper and back section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  Integral | 8.29 (3.262) | 0.52 (3.884)
  Trabecular | 36.05 (31.815) | -11.69 (37.721)
  Cortical | 2.17 (0.944) | -0.94 (1.129)

42. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Supero-posterior Cortical vBMD Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Week 52 + 30 days to Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therpay, and region. Supero-posterior is the upper and back section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
mg/cm^3 | 9.30 (4.287) | -4.92 (5.130)

43. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Supero-posterior Cortical Thickness Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: Cortical thickness (measured in millimeters) was measured by QCT. Percent change was calculated as (thickness at Week 52 + 30 days (or Week 76 + 30 days) minus thickness at Baseline)/thickness at Baseline x 100%
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, n=32, 35 | -20.48 (3.614) | 1.00 (3.986)
  Week 76 + 30 days, n=31,30 | -3.52 (3.674) | -1.50 (4.423)

44. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Supero-posterior Cortical Thickness Via QCT at Week 76 + 30 Days
Description: Cortical thickness was measured by QCT. Change from baseline was calculated as thickness at Week 76 + 30 days minus thickness at Baseline.
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
millimeters | -0.95 (0.0537) | -0.067 (0.0647)

45. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Supero-posterior Cortical Thickness Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: Cortical thickness (measured in millimeters) was measured by QCT. Percent change was calculated as (thickness at Week 76 + 30 days minus thickness at Week 52 + 30 days)/thickness at Week 52 + 30 days x 100%.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change | 32.42 (10.358) | -7.80 (2.383)

46. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Supero-posterior Cortical Thickness Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: Cortical thickness was measured by QCT. Change was calculated as thickness at Week 76 + 30 days minus thickness at Week 52 + 30 days.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
millimeters | 0.18 (0.049) | -0.05 (0.059)

47. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Supero-anterior Integral, Trabecular, and Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 daysor Week 76 + 30 days was calculated as (vBMD at Week 52 + 30 days(or Week 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Supero-anterior is the upper and front section of the FN.
Time Frame: Baseline, Week 52 plus 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -6.56 (2.106) | -0.58 (2.311)
  Week 52 + 30 days, Trabecular, n=32, 35 | 3.59 (4.719) | 2.82 (5.180)
  Week 52 + 30 days, Cortical, n=32, 35 | -1.91 (0.901) | -0.25 (0.977)
  Week 76 + 30 days, Integral, n=31, 30 | -4.97 (2.384) | -2.45 (2.838)
  Week 76 + 30 days, Trabecular, n=31, 30 | -0.85 (6.050) | 3.98 (7.171)
  Week 76 + 30 days, Cortical, n=31, 30 | -0.93 (0.745) | -1.49 (0.876)

48. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Supero-anterior Cortical vBMD Via QCT at Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Baseline at Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at baseline and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Supero-anterior is the upper and front section of the FN.
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
mg/cm^3 | -4.555 (3.5006) | -7.553 (4.1177)

49. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Supero-anterior Integral, Trabecular, and Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/vBMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Supero-anterior is the upper and front section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  Integral | 2.96 (2.202) | -1.81 (2.609)
  Trabecular | -2.78 (4.677) | 6.63 (5.531)
  Cortical | 1.19 (0.778) | -1.28 (0.912)

50. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Supero-anterior Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Week 52 + 30 days to Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Supero-anterior is the upper and front section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
mg/cm^3 | 5.19 (3.686) | -6.24 (4.319)

51. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Supero-anterior Cortical Thickness Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: Cortical thickness (measured in millimeters) was measured by QCT. Percent change was calculated as (thickness at Week 52 + 30 days(or Week 76 + 30 days) minus thickness at Baseline)/thickness at Baseline x 100%.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, n=32, 35 | -13.45 (5.002) | 5.05 (5.453)
  Week 76 + 30 days, n=31, 30 | -4.23 (4.491) | -4.78 (5.327)

52. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Supero-anterior Cortical Thickness Via QCT at Week 76 + 30 Days
Description: as for outcome 44
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
millimeters | -0.117 (0.0484) | -0.087 (0.0575)

53. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Supero-anterior Cortical Thickness Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: as for outcome 45
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change | 14.02 (6.779) | -13.65 (7.995)

54. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Supero-anterior Cortical Thickness Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: as for outcome 46
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
millimeters | 0.11 (0.052) | -0.13 (0.061)

55. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Infero-posterior Integral, Trabecular, and Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 days or Week 76 + 30 days was calculated as (vBMD at Week 52 + 30 days (or Week 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-posterior is the lower and back section of the FN.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -4.11 (1.074) | 1.74 (1.200)
  Week 52 + 30 days, Trabecular, n=32, 35 | -84.08 (270.700) | 282.16 (297.445)
  Week 52 + 30 days, Cortical, n=32, 35 | -3.42 (1.531) | 1.14 (1.694)
  Week 76 + 30 days, Integral, n=31, 30 | -3.11 (0.933) | 0.01 (1.147)
  Week 76 + 30 days, Trabecular, n=31, 30 | 24.46 (17.473) | 13.54 (20.790)
  Week 76 + 30 days, Cortical, n=31, 30 | -1.32 (1.234) | -1.17 (1.492)

56. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Infero-posterior Cortical vBMD Via QCT at Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Baseline at Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at baseline and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-posterior is the lower and back section of the FN.
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
mg/cm^3 | -12.424 (8.9945) | -10.244 (10.8703)

57. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Infero-posterior Integral, Trabecular, and Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/vBMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-posterior is the lower and back section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  Integral | 1.47 (1.183) | -1.87 (1.435)
  Trabecular | -39.81 (130.071) | 161.81 (154.179)
  Cortical | 2.67 (1.728) | -2.50 (2.076)

58. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Infero-posterior Cortical vBMD Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Week 52 + 30 days to Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-posterior is the lower and back section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
mg/cm^3 | 15.48 (11.544) | -17.59 (13.865)

59. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Infero-posterior Cortical Thickness Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: as for outcome 43
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 39
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, n=32, 35 | 0.47 (1.977) | -1.27 (2.180)
  Week 76 + 30 days, n=31, 30 | -1.46 (1.593) | -0.11 (1.910)

60. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Infero-posterior Cortical Thickness Via QCT at Week 76 + 30 Days
Description: as for outcome 44
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
millimeters | -0.082 (0.0816) | -0.048 (0.0978)

61. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Infero-posterior Cortical Thickness Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: as for outcome 45
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change | -1.48 (1.552) | 2.04 (1.846)

62. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Infero-posterior Cortical Thickness Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: as for outcome 46
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
millimeters | -0.08 (0.078) | 0.07 (0.093)

63. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Infero-anterior Integral, Trabecular, and Cortical vBMD Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Baseline at Week 52 + 30 days or Week 76 + 30 days was calculated as (vBMD at Week 52 + 30 days (orWeek 76 + 30 days) minus vBMD at baseline)/vBMD at Baseline x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-anterior is the lower and front section of the FN.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, Integral, n=32, 35 | -4.35 (1.950) | 1.26 (2.163)
  Week 52, Trabecular, n=32, 35 | -161.59 (774.589) | 930.71 (851.727)
  Week 52, Cortical, n=32, 35 | -1.85 (1.309) | 0.85 (1.563)
  Week 76 + 30 days, Integral, n=31, 30 | -0.29 (2.301) | 0.54 (2.810)
  Week 76 + 30 days, Trabecular, n=31, 30 | 81.29 (35.959) | 37.81 (42.791)
  Week 76 + 30 days, Cortical, n=31, 30 | 1.45 (1.149) | -0.63 (1.409)

64. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Infero-anterior Cortical vBMD Via QCT at Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Baseline at Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at baseline and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-anterior is the lower and front section of the FN.
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
mg/cm^3 | 7.901 (6.9912) | -5.025 (8.5722)

65. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Infero-anterior Integral, Trabecular, and Cortical vBMD Via QCT From Week 52+30 Days to Week 76 + 30 Days
Description: vBMD (measured in milligrams per centimeters cubed [mg/cm^3]) was measured by QCT. Percent change from Week 52 + 30 days to Week 76 + 30 days was calculated as (vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days)/vBMD at Week 52 + 30 days x 100% and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-anterior is the lower and front section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change
  Integral | 5.05 (1.878) | 0.38 (2.268)
  Trabecular | -90.60 (167.792) | 260.13 (199.323)
  Cortical | 3.68 (1.649) | -1.64 (2.016)

66. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Infero-anterior Cortical vBMD Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: vBMD was measured by QCT. Change from Week 52 + 30 days to Week 76 + 30 days was calculated as vBMD at Week 76 + 30 days minus vBMD at Week 52 + 30 days and was assessed by an analysis of covariance (ANCOVA) with terms for treatment, baseline value, prior therapy, and region. Infero-anterior is the lower and front section of the FN.
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
mg/cm^3 | 20.15 (9.677) | -10.73 (11.830)

67. Post Hoc Outcome: Adjusted Percent Change From Baseline in Femoral Neck (FN) Infero-anterior Cortical Thickness Via QCT at Week 52 + 30 Days and Week 76 + 30 Days
Description: Cortical thickness (measured in millimeters) was measured by QCT. Percent change was calculated as (thickness at Week 52 + 30 days (orWeek 76 + 30 days) minus thickness at Baseline)/thickness at Baseline x 100%.
Time Frame: Baseline, Week 52 + 30 days, and Week 76 + 30 days
Population: as for outcome 27
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 32 | 35
percent change
  Week 52 + 30 days, n=32, 35 | -6.05 (2.393) | 0.64 (2.656)
  Week 76 + 30 days, n=31, 30 | -3.59 (2.804) | 0.39 (3.421)

68. Post Hoc Outcome: Adjusted Change From Baseline in Femoral Neck (FN) Infero-anterior Cortical Thickness Via QCT at Week 76 + 30 Days
Description: Cortical thickness was measured by QCT. Change was calculated as thickness at Week 76 + 30 days minus thickness at Baseline.
Time Frame: Baseline and Week 76 + 30 days
Population: as for outcome 40
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 31 | 30
millimeters | -0.120 (0.0931) | -0.040 (0.1135)

69. Post Hoc Outcome: Adjusted Percent Change in Femoral Neck (FN) Infero-anterior Cortical Thickness Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: as for outcome 45
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
percent change | 3.12 (2.127) | 1.56 (2.257)

70. Post Hoc Outcome: Adjusted Change in Femoral Neck (FN) Infero-anterior Cortical Thickness Via QCT From Week 52 + 30 Days to Week 76 + 30 Days
Description: as for outcome 46
Time Frame: Week 52 + 30 days and Week 76 + 30 days
Population: as for outcome 28
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 30 | 30
millimeters | 0.09 (0.065) | 0.01 (0.078)

71. Post Hoc Outcome: Adjusted Change From Baseline in Albumin-adjusted Serum Calcium (AASC) at Week 52 and Week 76
Description: AASC levels were measured from blood samples. AASC is the amount of free calcium circulating in the blood and calcium is required for good bone health. Change from baseline was calculated as the Week 52or Week 76 value minus the baseline value and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Baseline, Week 52, and Week 76
Population: as for outcome 7
Measure: Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 73 | 83
millimoles per Liter (mmol/L)
  Week 52, n=73, 83 | 0.01 (0.009) | 0.03 (0.009)
  Week 76, n=64, 75 | 0.03 (0.010) | 0.04 (0.010)

72. Post Hoc Outcome: Adjusted Change in Albumin-adjusted Serum Calcium (AASC) From Week 52 to Week 76
Description: AASC levels were measured from blood samples. AASC is the amount of free calcium circulating in the blood and calcium is required for good bone health. Change from Week 52 was calculated as the Week 76 value minus the Week 52 value and was assessed by an ANCOVA with terms for treatment, baseline value, prior therapy, and region.
Time Frame: Week 52 and Week 76
Population: as for outcome 10
Measure: Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Arm/Group | Rosiglitazone in DB Period; Metformin in OL Period | Metformin in DB Period; Metformin in OL Period
Number analyzed (Participants) | 64 | 74
millimoles per Liter (mmol/L) | 0.01 (0.011) | 0.00 (0.010)

ADVERSE EVENTS:
Time Frame: 76 weeks
Description: Serious adverse events (SAEs) and AEs were collected in the Safety Population, comprised of all randomized participants who received at least one dose of study medication.
Groups:
- Rosiglitazone: DB: Rosiglitazone (RSG) initiated at a total daily dose of 4 milligrams (mg). RSG could be uptitrated to a total daily dose of 8 mg at Week 4 in the 52-week Double-Blind (DB) Period.
- Metformin: DB: Metformin (MET) initiated at a total daily dose of 1000 mg. MET could be uptitrated to 1500 mg/day at Week 2 and to 2000 mg/day at Week 4 in the 52-week DB Period.
- Rosiglitazone: MET OL: At Week 52, all participants receiving RSG in the DB Period were switched to open-label Metformin (MET) therapy for 24 weeks during the Open-label (OL) Period; all participants were force-titrated from 1000 mg/day to 2000 mg/day over a 4-week period. However, participants could be down-titrated to alleviate any MET-related tolerability issues.
- Metformin: MET OL: At Week 52, all participants receiving MET in the DB Period were switched to open-label MET therapy for 24 weeks during the OL Period; all participants were force-titrated from 1000 mg/day to 2000 mg/day over a 4-week period. However, participants could be down-titrated to alleviate any MET-related tolerability issues.
Arm/Group | Rosiglitazone: DB | Metformin: DB | Rosiglitazone: MET OL | Metformin: MET OL
Serious Adverse Events (participants affected / at risk) | 7/114 | 5/111 | 0/76 | 0/84
Other Adverse Events (participants affected / at risk) | 47/115 | 45/111 | 12/76 | 8/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone: DB (N=114) | Metformin: DB (N=111) | Rosiglitazone: MET OL (N=76) | Metformin: MET OL (N=84)
Device dislocation (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone: DB (N=115) | Metformin: DB (N=111) | Rosiglitazone: MET OL (N=76) | Metformin: MET OL (N=84)
Diarrhoea (Gastrointestinal disorders) | 3 | 15 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 6 | 0 | 0
Oedemal peripheral (General disorders) | 17 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 7 | 1 | 0
Influenza (Infections and infestations) | 3 | 6 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1 | 0
Headache (Nervous system disorders) | 9 | 5 | 1 | 1
Weight increased (Investigations) | 9 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.